CLINICAL TRIAL: NCT02581553
Title: A Phase 1, Randomized, Open-Label, Crossover Study to Assess the Relative Bioavailability of Lesinurad/Allopurinol Fixed Dose Combination Tablets and Coadministered Lesinurad and Allopurinol Tablets and the Effect of Food on the Pharmacokinetics of Lesinurad/Allopurinol Fixed Dose Combination Tablets in Healthy Adult Male Subjects
Brief Title: Lesinurad/Allopurinol 200/300 FDC Tablets Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RDEA594-501
Record Dates: First submitted 2015-10-12; First posted 2015-10-21 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence AB (Experimental): Day 1: lesinurad/allopurinol FDC tablets (Treatment A); Day 8: lesinurad + allopurinol (Treatment B)
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence BA (Experimental): Day 1: lesinurad + allopurinol (Treatment B); Day 8: lesinurad/allopurinol FDC tablets (Treatment A).
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence CD (Experimental): Day 1: lesinurad/allopurinol FDC tablets (Treatment C [fasted]); Day 8: lesinurad/allopurinol FDC tablets (Treatment D [fed]).
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets
- Sequence DC (Experimental): Day 1: lesinurad/allopurinol FDC tablets (Treatment D [fed]); Day 8: lesinurad/allopurinol FDC tablets (Treatment C [fasted]).
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablets
- Sequence EF (Experimental): Day 1: lesinurad/allopurinol 200/200 FDC tablets (Treatment E); Day 8: coadministered lesinurad 200 mg + allopurinol 200 mg (100 mg × 2)
  Interventions: Drug: lesinurad 200 mg; Drug: lesinurad/allopurinol 200/200 FDC tablets; Drug: allopurinol 200 mg
- Sequence FE (Experimental): Day 1: coadministered lesinurad 200 mg + allopurinol 200 mg (100 mg × 2) (Treatment F); Day 8: lesinurad/allopurinol 200/200 FDC tablets (Treatment E).
  Interventions: Drug: lesinurad 200 mg; Drug: lesinurad/allopurinol 200/200 FDC tablets; Drug: allopurinol 200 mg

INTERVENTIONS:
Drug: lesinurad/allopurinol 200/300 FDC tablets
  Arms: Sequence AB; Sequence BA; Sequence CD; Sequence DC
Drug: lesinurad 200 mg
  Arms: Sequence AB; Sequence BA; Sequence EF; Sequence FE
Drug: allopurinol 300 mg
  Arms: Sequence AB; Sequence BA
Drug: lesinurad/allopurinol 200/200 FDC tablets
  Arms: Sequence EF; Sequence FE
Drug: allopurinol 200 mg
  Arms: Sequence EF; Sequence FE

SUMMARY:
This study will assess relative bioavailability of lesinurad/allopurinol fixed dose combination (FDC), its individual components and the effect of food.

DETAILED DESCRIPTION:
The study comprises 2 parts. Part 1 will assess the relative BA of lesinurad/allopurinol FDC and monocomponents in fasted subjects. Part 2 will assess the effect of food on the PK of FDC tablets.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ranging between 18 kg/m2 and 40 kg/m2.
* Screening serum urate level is ≤ 7.0 mg/dL.

Exclusion Criteria:

* Asian subject who has a positive test for the HLA-B*5801 allele.
* History or suspicion of kidney stones.
* Estimated creatinine clearance, as determined at Screening, of < 90 mL/min calculated by the Cockcroft-Gault formula using ideal body weight.
* Undergone major surgery within 3 months prior to Screening.
* Donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1or has given a plasma donation within 4 weeks prior to Day 1.
* Inadequate venous access or unsuitable veins for repeated venipuncture.
* Received any strong or moderate enzyme-inducing drug or product within 2 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) endpoints in terms of maximum observed concentration (Cmax) for lesinurad/allopurinol 200/300 and 200/200 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Days 1 and Day 8
  Cmax is the maximum observed concentration of a drug after administration
PK endpoints in terms of time of occurrence of maximum observed concentration (tmax) for lesinurad/allopurinol 200/300 and 200/200 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Day 1 and Day 8
  Tmax is the time of occurrence of cmax
PK endpoints in terms of area under the plasma concentration time curve from zero to the last quantifiable sampling timepoint (AUC last) for lesinurad/allopurinol 200/300 and 200/200 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Day 1 and Day 8
  AUC last is the area under the plasma concentration time curve from zero to the last quantifiable sampling timepoint
PK endpoints in terms of area under the plasma concentration time curve from and from zero to infinity (AUC 0-∞) for lesinurad/allopurinol 200/300 and 200/200 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Day 1 and Day 8
  AUC 0-∞ is a meausre of total concentration from time zero to infinity
PK endpoints in terms of apparent terminal half-life (t1/2) for lesinurad/allopurinol 200/300 and 200/200 FDC tablets relative to lesinurad and allopurinol monocomponent tablets | Day 1 and Day 8
  t1/2 is a measure of apparent terminal half-life

SECONDARY OUTCOMES:
Incidence of Adverse Events in terms of changes in laboratory parameters | 6 weeks
Incidence of Adverse Events in terms of electrocardiogram parameters | 6 weeks
Incidence of Adverse Events in terms of vital signs | 6 weeks
Incidence of Adverse Events in terms of physical examination findings | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: N. Bhakta, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Austin, Texas, United States